CLINICAL TRIAL: NCT02855788
Title: Phase II Study of Metronomic Chemotherapy Using POLF Regimen in the Treatment of Advanced Gastric Cancer
Brief Title: Metronomic Chemotherapy in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Seattle Integrative Cancer Center (Unknown)
Responsible Party: Principal Investigator, Nick Chen, Visiting Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2016-206
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Metastatic Gastric Cancer; Locally Advanced Gastric Cancer
Keywords: gastric cancer; gastroesophageal cancer; metastatic; advanced
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POLF regimen (Experimental): Paclitaxel 60mg/m2, Oxaliplatin 50mg/m2, Leucovorin 20mg/m2, and 5-FU 425mg/m2 IV weekly
  Interventions: Drug: Paclitaxel 60mg/m2, Oxaliplatin 50mg/m2, Leucovorin 20mg/m2, and 5-FU 425mg/m2 IV weekly

INTERVENTIONS:
Drug: Paclitaxel 60mg/m2, Oxaliplatin 50mg/m2, Leucovorin 20mg/m2, and 5-FU 425mg/m2 IV weekly — metronomic chemotherapy
  Other Names: Taxol, Eloxatin

SUMMARY:
phase II study of weekly metronomic chemotherapy using weekly Paclitaxel, Oxaliplatin, Leucovorin and 5-FU (POLF) in patients with advanced gastric cancer

DETAILED DESCRIPTION:
About 80% of patients with advanced gastric cancer are diagnosed at an advanced stage with limited treatment options including systemic chemotherapy with or without radiation. Commonly used maximally tolerated dose (MTD) chemotherapy such as DCT, ECF, FOLFOX regimens induce responses in the range of 20 to 50% with median survival in the range of 10 to 12 months. Metronomic chemotherapy has been found to have more consistent anti-tumor effects through anti-angiogenic and immunomodulating effects. Preliminary clinical studies of weekly POLF have found very encouraging clinical activities and low overall toxicities in pancreatic cancer and gastric cancer. Here we conduct a formal clinical trial to determine the clinical efficacy and side effect profiles of this regimen in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed gastric cancer AJCC stage III or IV
2. measurable disease based on CT or endoscopy exam
3. non-surgical candidates or patients who declined surgery
4. non-radiation candidates or patients who declined radiation
5. patients who are able to sign informed consent
6. patients who are 2 weeks out and recovered from surgery
7. patients who have completed radiation to relieve obstructive symptoms
8. patient who previously received Oxaliplatin and 5-FU in other MTD regimens
9. adequate marrow function: neutrophil >1000/ul, Hgb >10g/dl, Plt>50,000

Exclusion Criteria:

1. allergic to any of the drugs involved
2. concurrent malignancies
3. severe co-morbidities of heart, lungs, kidneys and bone marrow
4. severe psychological disorder
5. severe malnutrition
6. difficult to heal or unhealed wound
7. ECOG performance status equal or over 3
8. uncontrolled complications from the malignancy
9. uncontrolled CNS metastasis
10. peripheral neuropathy grade 3 or above
11. pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-07 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
response rate | 3 months
  based on Recist 1.1

SECONDARY OUTCOMES:
adverse events | 2 years
  based on NCI-CTC v.2
progression free survival | 2 years
  median
overall survival | 2 years
  median

CONTACTS AND LOCATIONS:
Overall Officials: Jie Liu, M.D., Principal Investigator — Huashan Hospital; Nick N Chen, M.D., Ph.D., Principal Investigator — Seattle Integrative Cancer Center; Jun Zhang, M.D., Study Director — Huashan Hospital; Zhongguang Luo, M.D., Study Director — Huashan Hospital
Locations (2):
- Seattle Integrative Cancer Center, Seattle, Washington, United States
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes